CLINICAL TRIAL: NCT06408545
Title: Acceptance and Commitment Therapy for Problematic Chemsex: a Pilot Study
Brief Title: Acceptance and Commitment Therapy for Problematic Chemsex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Apoyo Positivo (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-324
Record Dates: First submitted 2024-04-22; First posted 2024-05-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-04

CONDITIONS: Hypersexuality; Compulsive Sexual Behavior; Sexualized Drug Use (Chemsex)
Keywords: Sexuality; Risky sexual behavior
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder; Chemsex; Sexuality | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT group (Experimental): 8 individual weekly sessions including ACT methods
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Acceptance and Commitment Therapy methods were focused on promoting Values clarification, Acceptance, Cognitive defusion, Committed action and Flexible attention to the present moment, and included methods such as the Garden Metaphor, Funeral exercise or Mindfulness training.

SUMMARY:
Investigation of the efficacy of Acceptance and Commitment Therapy (ACT) for the psychological treatment of problematic chemsex. As a pilot study, the intervention will be tested in a small group.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will be assessed to determine eligibility for study entry.

Patients who meet eligibility requirements will receive psychological intervention consisting in an 8-session individual on line-delivered ACT-based treatment.

The participants will be assessed through self-report instruments before and after treatment and at 3 months follow-up.

The pilot study will not include a control group.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years-old
* Spanish speaking
* having used psychoactive substances to facilitate, maintain and/or improve sexual relations in the last year
* significant score on the HBI Inventory (of 53 or more)
* clinically significant discomfort related to sexual practices
* degree of interference in his/her life of sexual practices greater than or equal to 5 out of 10
* desire to improve/reduce excessive sexual behaviour

Exclusion Criteria:

* receiving psychological or psychopharmacological treatment
* intellectual disability
* substance dependence (use not associated with sex)
* personality disorder or other serious or chronic mental disorder diagnosed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Hypersexual Behavior Inventory (HBI) | Change from Baseline Hypersexuality at 5 months
  The Hypersexual Behavior Inventory is a 19-item, seven-point Likert-type scale. Scores range between 19 and 95. Higher scores indicate higher levels of Hypersexuality and worse outcome. The presence of a problem of hypersexuality is considered when the score is equal or higher than 53.

SECONDARY OUTCOMES:
Change in Drug Abuse Screening Test (Dast-10) | Change from Baseline Drug Abuse at 5 months
  Drug Abuse Screening Test is a self-administered 10-item questionnaire with dichotomous (Yes/No) responses designed to identify individuals with problematic drug use. Scores range between 0 and 10. Different cutoff points are established regarding problematic substance use, as follows: 0 = low risk or abstinence, 1-2 = risk, 3-5 = harmful, > 6 = substance dependence. The presence of a problem of substance abuse is considered when the score is equal or higher than 3.
Change in Brief Symptom Inventory (BSI) | Change from Baseline Anxiety and Depression at 5 months
  Anxiety and Depression subscales of The Brief Symptom Inventory (BSI) include 15 items, each item is rated on a 5-point scale (0 to 4) according to manifestations of anxiety and depression symptoms in the last 30 days (ranging from ''not at-all'' to ''extremely''). Higher scores indicate higher levels of anxiety and depression and worse outcome.
Change in Acceptance and Action Questionnaire (AAQ-II) | Change from Baseline psychological inflexibility at 5 months
  Acceptance and Action Questionnaire assesses psychological inflexibility. It is a 7-item, seven-point Likert-type scale. Scores range between 7 and 49. Higher scores indicate higher levels of psychological inflexibility and worse outcome. The presence of a problem of psychological inflexibility is considered when the score is equal or higher than 27.
Change in Short Internalized Homonegativity Scale (SIHS) | Change from Baseline Internalized Homonegativity at 5 months
  Internalized homophobia has been defined as "the internalization of society's homophobic attitudes within a lesbian, gay, or bisexual individual". The Short Internalized Homonegativity Scale measures this phenomenon through a 13-item, five-point Likert-type scale ranging from strongly disagree to strongly agree. Scores range between 13 and 65. Higher scores indicate higher levels of internalized homonegativity and worse outcome. For men, the mean total score is 28.16 (SD = 8.23). The questionnaire includes three sub-scales: public identification as homosexual, sexual comfort with homosexual and social comfort with homosexual people.
Change in Social and Emotional Loneliness in Adults (SESLA) | Change from Baseline Emotional Loneliness at 5 months
  The Scale of Evaluation of Social and Emotional Loneliness in Adults evaluates loneliness. The scale is comprised of 3 factors: social loneliness, which reflects the lack of friends and social relationships, family loneliness, which reflects the lack of a supportive family environment for the person, and romantic loneliness, which reflects the lack of an intimate romantic relationship. The scale consists of 15 items with which agreement or disagreement is shown according to a 7-point Likert-type scale. Scores range between 15 and 105. Higher scores indicate higher levels of loneliness and worse outcome.
Change in Awareness, Courage and Responsiveness Scale (ACRS) | Change from Baseline Awareness, Courage and Responsiveness at 5 months
  The Awareness, Courage and Responsiveness Scale is the first measure created to assess a contextual-behavioral model of Intimacy, rooted in the Functional Analytic Psychotherapy. It is a 24-item self-report assessment to evaluate the components of the ACR model, using a 7-point Likert-type scale from 1 (never true) to 7 (always true). The scale is comprised of 4 subscales: Others-Awareness (OA), 5 items; Self-Awareness (SA), 6 items; Courage (C), 6 items; and Responsiveness (R), 7 items. The total sum of the items of the scale is considered a global measure of Intimacy (ACRS-T). Scores range between 24 and 168. Higher scores indicate higher levels of skills to generate intimacy and better outcome.
Change in The Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT) | Change from Baseline psychological flexibility at 5 months
  The Comprehensive Assessment of Acceptance and Commitment Therapy Processes Change is a 23-item, seven-point Likert-type scale. Scores range between 0 and 138. Higher scores indicate higher levels of psychological flexibility and better outcome. This scale provides more accurate information about each of the psychological processes underlying psychological flexibility. Specifically, it consists of 3 subscales: openness, awareness, and action.
Change in the Life Values Questionnaire (VLQ) | Change from Baseline value consistency living at 5 months
  The Life Values Questionnaire relates to 10 domains of different life values, which include: family, marriage/intimate partner relationships, parenthood, friendship, work, education, leisure, spirituality, citizenship, and physical self-care. Participants are asked to evaluate on a Likert scale from 0 to 10 the degree of importance they give to these values, where 0 is of little importance and 10 is of great importance. Additionally, they are asked to rate the degree of consistency with which they engage in actions committed to these values, ranging from 0 to 10. Scores are obtained for different sub-scales: importance, consistency, and discrepancy. As a global score for the questionnaire, the composite score is obtained by subtracting the consistency score from the importance score. Higher scores in discrepancy indicates lower levels of value consistency living and worse outcome.
Change in Time spent planning or practicing sex per week | Through study completion, an average of 5 months
  Time spent (hours) planning or practicing sex during last week. Higher number of hours indicate worse outcome.
Change in Frequency of chemsex encounters per week | Through study completion, an average of 5 months
  Self-monitoring: Frequency of practicing chemsex during last week. Higher number of chemsex encounters indicate worse outcome.
Change in number of different sexual partners per week | Through study completion, an average of 5 months
  Self-monitoring: Number of different sexual partners during last week. Higher number of different sexual partners indicate worse outcome.
Change in Frequency of substance consumption per week | Through study completion, an average of 5 months
  Self-monitoring: Frequency of consuming substances during last week. Higher number of substances consumed indicate worse outcome.
Change in Frequency of risky sexual practices per week | Through study completion, an average of 5 months
  Self-monitoring: Frequency of risky sexual practices during the last week. Higher number of risky sexual practices indicate worse outcome.
Change in number of new diagnoses of sexually transmitted infections per week | Through study completion, an average of 5 months
  Self-monitoring: Number of new diagnoses of sexually transmitted infections. Higher number of new diagnoses indicate worse outcome.
Change in Intensity of cravings subjective scale | Through study completion, an average of 5 months
  Global self-assessment of intensity of cravings Visual Analogue Scale-ratings. Scores range from 0 = very low intensity to 10 = very high intensity. Higher scores indicate higher levels of intensity of cravings and worse outcome
Change in Interference of cravings subjective scale | Through study completion, an average of 5 months
  Global self-assessment of interference of cravings Visual Analogue Scale-ratings. Scores range from 0 = very low interference to 10 = very high interference. Higher scores indicate higher levels of interference of cravings and worse outcome.
Change in Frequency of value committed actions per week | Through study completion, an average of 5 months
  Self-monitoring: Frequency of value committed actions in presence of craving during last week. Higher number of value committed actions indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Montesinos, Ph.D., Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT06408545/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT06408545/ICF_001.pdf